CLINICAL TRIAL: NCT04783415
Title: A Phase II Study of BTK Inhibitor Acalabrutinib and PI3Kδ Inhibitor Umbralisib in Combination With Ublituximab (AU2) in Patients With Previously Untreated Mantle Cell Lymphoma (MCL)
Brief Title: Acalabrutinib, Umbralisib, and Ublituximab for the Treatment of Previously Untreated Mantle Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20459; NCI-2021-00498 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20459 (Other: City of Hope Comprehensive Cancer Center); P30CA033572 (NIH)
Record Dates: First submitted 2021-02-25; First posted 2021-03-05 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — acalabrutinib; ublituximab; LFB-R603; umbralisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (ublituximab, acalabrutinib, umbralisib) (Experimental): Patients receive ublituximab IV over 90 minutes-4 hours on days 1, 8, and 15 of cycle 1 and days 1 of cycles 2-6. Patients also receive acalabrutinib PO BID and umbralisib PO QD on days 1-28. Treatment repeats every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients receive ublituximab IV on day 1 on cycles 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30. Patients also receive acalabrutinib Po BID and umbralisib PO QD on day 1-28. Treatment repeats every 28 days for 24 cycles in the absence of disease progression of unacceptable toxicity.
  Interventions: Drug: Acalabrutinib; Biological: Ublituximab; Drug: Umbralisib

INTERVENTIONS:
Drug: Acalabrutinib — Given PO
  Other Names: ACP-196; Bruton Tyrosine Kinase Inhibitor ACP-196; Calquence
Biological: Ublituximab — Given IV
  Other Names: LFB-R603; TG-1101; TG-20; TGTX-1101
Drug: Umbralisib — Given PO
  Other Names: 2-((1S)-1-(4-Amino-3-(3-fluoro-4-(1-methylethoxy)phenyl)-1H-pyrazolo(3,4-d)pyrimidin-1-yl)ethyl)-6-fluoro-3-(3-fluorophenyl)-4H-1-benzopyran-4-one; RP-5264; RP5264; TGR-1202

SUMMARY:
This phase II trial studies the effects of acalabrutinib, umbralisib, and ublituximab in treating previously untreated mantle cell lymphoma. Acalabrutinib and umbralisib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Ublituximab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. Giving acalabrutinib and umbralisib with ublituximab may work better in treating mantle cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the anti-tumor activity of acalabrutinib, umbralisib and ublituximab (AU2) regimen as induction therapy in patients with treatment-naïve mantle cell lymphoma (MCL), as assessed by the complete response (CR) rate.

SECONDARY OBJECTIVES:

I. Evaluate the overall response rate (ORR) to AU2 in treatment-naive MCL. II. Evaluate the progression-free survival (PFS), overall survival (OS) and duration of response (DOR) in patients with treatment-naïve MCL who received AU2.

III. Evaluate the safety and tolerability of AU2 in patients with treatment-naive MCL.

EXPLORATORY OBJECTIVES:

I. Examine the T-cell populations and functionality in patients treated with AU2.

II. Explore the predictive value of minimal residual disease (MRD) in MCL. III. Explore the mechanisms of resistance to AU2 therapy.

OUTLINE:

INDUCTION: Patients receive ublituximab intravenously (IV) over 90 minutes-4 hours on days 1, 8, and 15 of cycle 1 and days 1 of cycles 2-6. Patients also receive acalabrutinib orally (PO) twice daily (BID) and umbralisib PO once daily (QD) on days 1-28. Treatment repeats every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive ublituximab IV on day 1 on cycles 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30. Patients also receive acalabrutinib Po BID and umbralisib PO QD on day 1-28. Treatment repeats every 28 days for 24 cycles in the absence of disease progression of unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Histologically confirmed mantle cell lymphoma with documentation of monoclonal CD20+ B cells that have a chromosome translocation t(11;14)(q13;q32) and/or overexpress cyclin D1
* Age >= 65 years; or >= 50 years and deemed ineligible for aggressive induction therapy or autologous stem cell transplant by the investigator, or unwilling to undergo aggressive induction; or >= 18 years with documented del(17p), or TP53 mutation, or complex karyotype (CK) by cytogenetics and/or fluorescence in situ hybridization (FISH) studies
* Requiring treatment for MCL, and for which no prior systemic anticancer therapies have been received (local radiotherapy not exceeding a total dose of 20 Gy at least 2 weeks prior the first dose of study therapy is allowed)
* Measurable disease by computed tomography (CT) or positron emission tomography (PET)/CT scan with one or more sites of disease >= 1.5 cm in longest dimension (including splenomegaly), or bone marrow involvement with or without malignant lymphocytosis
* Without bone marrow involvement: Absolute neutrophil count (ANC) >= 1000/mm^3

  * NOTE: Growth factor is not permitted within 7 days of ANC assessment unless cytopenia is secondary to disease involvement
* With bone marrow involvement: ANC >= 500/mm^3

  * NOTE: Growth factor is not permitted within 7 days of ANC assessment unless cytopenia is secondary to disease involvement
* Without bone marrow involvement: Platelets >= 75,000/mm^3

  * NOTE: Platelet transfusions are not permitted within 7 days of platelet assessment unless cytopenia is secondary to disease involvement
* With bone marrow involvement: Platelets >= 30,000/mm^3

  * NOTE: Platelet transfusions are not permitted within 7 days of platelet assessment unless cytopenia is secondary to disease involvement
* Total bilirubin =< 1.5 X upper limit of normal (ULN) or =< 3X ULN for Gilbert's disease
* Aspartate aminotransferase (AST) =< 2.5 x ULN
* Alanine aminotransferase (ALT) =< 2.5 x ULN
* Creatinine clearance of >= 30 mL/min per 24 hour urine test or the Cockcroft-Gault formula
* If not receiving anticoagulants: International normalized ratio (INR) OR prothrombin (PT) =< 1.5 x ULN. If on anticoagulant therapy: PT must be within therapeutic range of intended use of anticoagulants
* If not receiving anticoagulants: Activated partial thromboplastin time (aPTT) =< 1.5 x ULN. If on anticoagulant therapy: aPTT must be within therapeutic range of intended use of anticoagulants
* Left ventricular ejection fraction (LVEF) >= 40%
* Women of childbearing potential (WOCBP): negative serum pregnancy test
* Agreement by females and males of childbearing potential to use an highly effective method of birth control or abstain from heterosexual activity for the course of the study through at least 2 days after the last dose of acalabrutinib for females, and at least 4 months after the last dose of ublituximab or umbralisib, whichever comes later, for both men and women

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Chronic use of corticosteroids >= 20 mg/day (short-term use of steroids < 14 days is allowed)
* Major surgical procedure within 28 days of start of protocol therapy. Note: If a subject had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug
* Known history of hypersensitivity or anaphylaxis to study drug(s) including active product or excipient components
* Concurrent participation in another therapeutic clinical trial
* Subjects for whom the goal of therapy is tumor debulking before stem cell transplant
* History of prior malignancy. Exceptions include malignancy treated with curative intent and no known active disease present for >= 2 years prior to initiation of protocol therapy; adequately treated non-melanoma skin cancer or lentigo maligna (melanoma in situ) without evidence of disease; adequately treated in situ carcinomas (e.g., cervical, esophageal, etc.) without evidence of disease; asymptomatic prostate cancer managed with "watch and wait" strategy
* Uncontrolled AIHA (autoimmune hemolytic anemia) or ITP (idiopathic thrombocytopenic purpura)
* Requires treatment with proton pump inhibitors (e.g., omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole, or pantoprazole). Subjects receiving proton pump inhibitors who switch to H2-receptor antagonists or antacids are eligible for enrollment to this study
* Requires treatment with a strong cytochrome P450 3A4 (CYP3A4) inhibitor/inducer
* Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel that is likely to affect absorption, symptomatic inflammatory bowel disease, partial or complete bowel obstruction, or gastric restrictions and bariatric surgery, such as gastric bypass
* Presence of a gastrointestinal ulcer diagnosed by endoscopy within 3 months before screening
* Known bleeding disorders (e.g., von Willebrand's disease or hemophilia)
* History of significant cerebrovascular disease/event, including stroke, myocardial infarction or intracranial hemorrhage, within 6 months prior to start of protocol therapy
* Known active central nervous system (CNS) involvement by lymphoma, including leptomeningeal involvement
* Clinically significant cardiovascular disease such as symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any class III or IV cardiac disease as defined by the New York Heart Association Functional Classification. Note: Subjects with controlled, asymptomatic atrial fibrillation can enroll on study
* Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 6 months)
* History of or current progressive multifocal leukoencephalopathy (PML)
* Inability to swallow and retain an oral medication
* Clinically significant uncontrolled illness, including active infection requiring antibiotics
* Live virus vaccines within 4 weeks of start of protocol therapy or planned administration of live virus vaccines during ublituximab therapy
* Evidence of chronic active hepatitis B (HBV, not including patients with prior hepatitis B vaccination; or positive serum Hepatitis B antibody) or chronic active hepatitis C infection (HCV), or active cytomegalovirus (CMV). If hepatitis B virus core (HBc) antibody is positive, the subject must be evaluated for the presence of HBV deoxyribonucleic acid (DNA) by polymerase chain reaction (PCR). If HCV antibody is positive, the subject must be evaluated for the presence of HCV RNA by PCR. If the subject is CMV IgG or CMV IgM positive, the subject must be evaluated for the presence of CMV DNA by PCR. Subjects with positive HBc antibody and negative HBV DNA by PCR are eligible. Subjects with positive HCV antibody and negative HCV RNA by PCR are eligible. Subjects who are CMV IgG or CMV IgM positive but who are CMV DNA negative by PCR are eligible. Patients with a prior known history of hepatitis B and those with a positive anti-HBc with negative hepatitis B surface antigen (HBsAg) at screening must be able to receive antiviral agents effective against hepatitis B
* Known history of human immunodeficiency virus (HIV) infection
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2025-09-20 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Alexey V Danilov, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Ublituximab, Acalabrutinib, Umbralisib): Patients receive ublituximab IV over 90 minutes-4 hours on days 1, 8, and 15 of cycle 1 and days 1 of cycles 2-6. Patients also receive acalabrutinib PO BID and umbralisib PO QD on days 1-28. Treatment repeats every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients receive ublituximab IV on day 1 on cycles 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30. Patients also receive acalabrutinib Po BID and umbralisib PO QD on day 1-28. Treatment repeats every 28 days for 24 cycles in the absence of disease progression of unacceptable toxicity.
  Acalabrutinib: Given PO
  Ublituximab: Given IV
  Umbralisib: Given PO
Period: Overall Study
Arm/Group | Treatment (Ublituximab, Acalabrutinib, Umbralisib)
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Ublituximab, Acalabrutinib, Umbralisib)
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 70 [55 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR) Rate After Induction (Six Cycles)
Description: Defined as the proportion of response-evaluable participants that achieve a CR at the end of the induction therapy. CR rate after the induction therapy was estimated by the proportion of response-evaluable patients achieving CR after the induction therapy, along with the 95% exact binomial confidence interval.
Time Frame: Participants were assessed at the end of the induction therapy (24 weeks post-baseline). The induction therapy included six 28-day cycles of the study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Ublituximab, Acalabrutinib, Umbralisib)
Number analyzed (Participants) | 12
percentage of participants | 100

2. Secondary Outcome: Overall Response Rate (ORR)
Description: Defined as the proportion of response-evaluable participants that achieve a best response of either CR or partial response (PR) during protocol therapy. ORR rate after induction therapy was estimated by the proportion of response-evaluable patients achieving ORR after induction therapy, along with the 95% exact binomial confidence interval.
Time Frame: Participants were followed up to 24 months after the end of protocol therapy.
Reporting Status: Not Posted, anticipated posting 2025-09

ADVERSE EVENTS:
Time Frame: Adverse Events were monitored/assessed at each 28-day cycle treatment and up to 30 days at the end of the protocol therapy. Currently, patients received the study treatment up to 12 cycles. All-Cause Mortality was monitored/assessed up to 30 months from the start time of the initial treatment.
Arm/Group | Treatment (Ublituximab, Acalabrutinib, Umbralisib)
All-Cause Mortality (participants affected / at risk) | 1/12
Serious Adverse Events (participants affected / at risk) | 4/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ublituximab, Acalabrutinib, Umbralisib) (N=12)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Covid-19 (Infections and infestations) | 1 (1)
Meningitis (Infections and infestations) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ublituximab, Acalabrutinib, Umbralisib) (N=12)
Anemia (Blood and lymphatic system disorders) | 8 (13)
Palpitations (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 5 (5)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (7)
BELCHING (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 11 (30)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (2)
HEARTBURN (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
MILD CHEST DISCOMFORT (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (12)
Oral pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (13)
Chills (General disorders) | 2 (2)
Edema limbs (General disorders) | 3 (5)
Facial pain (General disorders) | 1 (2)
Fatigue (General disorders) | 5 (6)
Fever (General disorders) | 2 (3)
Flu like symptoms (General disorders) | 2 (2)
Malaise (General disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 2 (2)
Pain (General disorders) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2)
Allergic Conjunctivities (Infections and infestations) | 1 (1)
Eye infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Thrush (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 4 (5)
Infusion related reaction (Injury, poisoning and procedural complications) | 9 (12)
Alanine aminotransferase increased (Investigations) | 4 (11)
Alkaline phosphatase increased (Investigations) | 3 (6)
Aspartate aminotransferase increased (Investigations) | 8 (16)
Blood bilirubin increased (Investigations) | 1 (4)
Blood lactate dehydrogenase increased (Investigations) | 8 (10)
Creatinine increased (Investigations) | 4 (5)
Lymphocyte count decreased (Investigations) | 4 (7)
Lymphocyte count increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 4 (9)
Platelet count decreased (Investigations) | 7 (11)
Weight gain (Investigations) | 5 (5)
Weight loss (Investigations) | 5 (7)
White blood cell decreased (Investigations) | 5 (9)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (13)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 5 (5)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hyperphosphatemia (Metabolism and nutrition disorders) | 5 (6)
Hyperuricemia (Metabolism and nutrition disorders) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 9 (14)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 7 (13)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 4 (5)
Dysgeusia (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 7 (9)
Paresthesia (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Mania (Psychiatric disorders) | 1 (1)
Psychosis (Psychiatric disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Glucosuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (8)
dog bite (Social circumstances) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 9 (29)
Hypotension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-06): https://cdn.clinicaltrials.gov/large-docs/15/NCT04783415/Prot_SAP_000.pdf